CLINICAL TRIAL: NCT05661708
Title: Use of Chitosan Powder in Loop Electrosurgical Excision Procedure to Reduce Postoperative Complications: A Randomized Controlled Trial
Brief Title: Use of Chitosan Powder in Loop Electrosurgical Excision Procedure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, Medical Doctor - Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MUGLA-9
Record Dates: First submitted 2022-12-13; First posted 2022-12-22 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Vaginal Bleeding; Loop Electrosurgical Excision
MeSH Terms: conditions — Uterine Hemorrhage | interventions — Chitosan

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): LEEP was performed in an outpatient setting by a single resident physician (KG). A full blood count was taken (hematocrit 1). The procedure was designed according to colposcopic findings such as the type of transformation zone and position of the lesion. After positioning of the patient, 50 mg of lidocaine spray (5 pumps, 10 mg in each pump) was applied to the ectocervix, then 2 mL bupivacaine hydrochloride was injected submucosally using a 27-gauge needle tip at the 3, 6, 9, and 12 o'clock locations in the ectocervix. LEEP was performed as described in a previous trial. After the hemostasis that obtained using the ball electrode at a 40-W coagulation setting, the remaining cervical tissue was washed with 20 ccs of sterile saline to ensure no active bleeding from the cervical wound. An empty spray pump was used because we cannot find any identical powder for the placebo
- Chitosan (Experimental): LEEP was performed in an outpatient setting by a single resident physician (KG). A full blood count was taken (hematocrit 1). The procedure was designed according to colposcopic findings such as the type of transformation zone and position of the lesion. After positioning of the patient, 50 mg of lidocaine spray (5 pumps, 10 mg in each pump) was applied to the ectocervix, then 2 mL bupivacaine hydrochloride was injected submucosally using a 27-gauge needle tip at the 3, 6, 9, and 12 o'clock locations in the ectocervix. LEEP was performed as described in a previous trial. After the hemostasis that obtained using the ball electrode at a 40-W coagulation setting, the remaining cervical tissue was washed with 20 ccs of sterile saline to ensure no active bleeding from the cervical wound. The application of 3 or 4 pumps of chitosan powder was carried out into the wound bed by spray pump which was prepared by a nurse.
  Interventions: Drug: Chitosan

INTERVENTIONS:
Drug: Chitosan — Chitosan is a biodegradable, natural polyaminosaccharide with a nontoxic, non-allergenic, positively-charged polysaccharide derived from the deacetylation of chitin. Due to its molecular characteristics, chitosan has been used for improved hemostasis. Furthermore, chitosan has an antimicrobial and wound-healing effect
  Arms: Chitosan

SUMMARY:
Early treatment of cervical intraepithelial neoplasia (CIN) II-III gives rise to a decrease in the incidence of invasive cervical cancer. Though there is no obvious consensus from randomized studies as to the optimal management of CIN II-III, loop electrosurgical excision procedure (LEEP) is the most extensively used method because of its technical ease, inexpensive, steep learning curve, and low rate of complications.

In spite of these benefits, current literature suggests that some patients experience some complications such as postoperative vaginal bleeding, abnormal vaginal discharge, abdominal pain, and infection. These adversely affect the recovery period, increase patient anxiety, readmission to the hospital for further treatment and encumber patients' daily life. Postoperative vaginal bleeding (PVB) is one of the most common and unpleasant of these complications. Its incidence has been reported to vary between 2% to 78%.

Many different types of treatments have been applied to avert or diminish PVC such as the use of vasopressin, tranexamic acid, Monsel's solution, and local hemostats (e.g., TachoSil or Tisseel), but these attempts have failed to show precise benefits over routine clinical approaches. Chitosan is a biodegradable, natural polyaminosaccharide with a nontoxic, non-allergenic, positively-charged polysaccharide derived from the deacetylation of chitin. Due to its molecular characteristics, chitosan has been used for improved hemostasis. Furthermore, chitosan has an antimicrobial and wound-healing effect. The current literature concerning the influence of using chitosan after the LEEP is limited to only one trial. The authors of that study reported that using chitosan after the LEEP can reduce vaginal bleeding and enhancing wound healing. However, that study has some limitations. Therefore, investigators designed this randomized trial to assess the effect of local chitosan implementation on postoperative vaginal bleeding and wound healing in LEEP

ELIGIBILITY:
Inclusion Criteria:

* women were aged > 21 years old
* women were not pregnant
* women who were undergoing LEEP.

Exclusion Criteria:

* Women with pelvic infection
* Women with abnormal vaginal bleeding
* Women with coagulopathy
* Women with chronic pain syndromes
* Women with psychiatric disorders
* Women with the previous hysterectomy with removal of the cervix,
* Women with a history of cervical cancer
* Women who could not complete follow-up calls

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
median early postoperative blood loss | 6 hours
  early postoperative blood loss using the difference in hematocrit values after LEEP and 24 h after the procedure according to the following formula: estimated blood loss = estimated blood volume × (hematocrit 1 - hematocrit 2) / hematocrit 1, where the estimated blood volume in milliliters = body weight in kilograms × 85

SECONDARY OUTCOMES:
Wound healing score | 1-4 weeks
  The imagine J software program (https://imagej.net/ij/) was used to measure the area of wounds. In order to determine the rate of wound healing, the formula used is [(initial area of treatment wound - remaining wound area)/initial area of treatment wound] × 100%.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kemal Güngördük, Menteşe, Muğla
  - Mugla Sıtkı Kocman University Education and Research Hospital, Muğla

IPD SHARING:
Plan to Share IPD: No